CLINICAL TRIAL: NCT02098824
Title: Symptomatic Treatment of Vascular Cognitive Impairment
Acronym: STREAM-VCI
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Dr. Niels Prins, MD, PhD, MD, PhD, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Crossover | Masking: Triple
Other Study IDs: NL45933.029.13
Record Dates: First submitted 2014-03-14; First posted 2014-03-28 (Estimated); Last update posted 2016-05-02 (Estimated); Status verified 2016-04

CONDITIONS: Mild Cognitive Impairment (Vascular); Mild Cognitive Disorder (Vascular); Vascular Dementia
Keywords: vascular cognitive impairment; treatment; cerebrovascular lesions; memory impairment; executive dysfunction; neuronal networks; white matter tracts; monoaminergic systems; cholinergic systems; DTI; rs-fMRI
MeSH Terms: conditions — Cognitive Dysfunction; Neurocognitive Disorders; Dementia, Vascular; Memory Disorders | interventions — Galantamine; Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Galantamine (Active Comparator): Single administration of capsule containing 16 mg Galantamine
  Interventions: Drug: Galantamine
- Placebo (Placebo Comparator): Single oral administration of capsule containing placebo
  Interventions: Drug: Placebo
- Methylphenidate (Active Comparator): Single administration of capsule containing 10 mg Methylphenidate
  Interventions: Drug: Methylphenidate

INTERVENTIONS:
Drug: Galantamine — Single administration of capsule containing 16 mg of Galantamine
  Other Names: Reminyl
  Arms: Galantamine
Drug: Methylphenidate — Single administration of capsule containing 10 mg of Methylphenidate
  Other Names: Ritalin
  Arms: Methylphenidate
Drug: Placebo — Single administration of capsule containing placebo
  Arms: Placebo

SUMMARY:
Single center threeway double blind cross over trial investigating the pharmacological responsivity in patients with VCI using a challenge aimed at the monoaminergic and cholinergic neuronal systems

DETAILED DESCRIPTION:
Vascular Cognitive Impairment is an important cause of cognitive impairment and dementia. Till now, there are no approved symptomatic treatments for Vascular Cognitive Impairment. Research on novel pharmacological treatments that may reduce clinical symptoms in these patients is needed. Evidence suggests that executive dysfunction and memory impairment in Vascular Cognitive Impairment are caused by damage to monoaminergic and cholinergic neurotransmitter-systems, respectively.

However, patients with Vascular Cognitive Impairment form a clinically heterogeneous group, i.e. the extent to which executive function and memory are affected differs from patient to patient. Previous intervention studies have not taken this inter-patient variability into account. Individually tailored pharmacological interventions, aimed at the affected neurotransmitter systems, may ameliorate cognitive symptoms in patients with Vascular Cognitive Impairment. Using a pharmacological challenge, it is possible to detect individual sensitivity to specific pharmacological interventions. Furthermore, with the use of novel MRI techniques, it is possible to correlate the location and severity of cerebrovascular lesions to impaired structural and functional connectivity in each subject.

The investigators will recruit 30 patients with Vascular Cognitive Impairment (according to the criteria of the American Heart Association/American Stroke Association), at the Alzheimer Center of the VU University Medical Center and the Utrecht University Medical Center. They will also undergo MRI, including diffusion tensor imaging MRI (DTI)/'fiber tracking'; and resting state (RS) functional MRI (fMRI). In a double-blind, three-way, case cross over trial, the investigators will study the effects of methylphenidate on executive function and of galantamine on episodic memory function. During three separate visits, patients will receive the pharmacological interventions (placebo, methylphenidate, and galantamine) at the investigators Clinical Research Unit. Also, during a study day the investigators will collect blood samples at different timepoints.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients
* Objective executive dysfunction and/or memory impairment on neuropsychological tests and imaging evidence of cerebrovascular disease (white matter changes (Fazekas ≥2, (lacunar) infarcts)
* Mini Mental State Examination (MMSE) ≥16
* Clinical Dementia Rating Score (CDR of 0.5-1)
* No contraindication for treatment with a Cholinesterase inhibitor (CEI) or Methylphenidate (MPH) (www.fk.cvz.nl)
* Assessed by the treating neurologist as mentally capable of understanding the implications of study participation
* Presence of an informant/caregiver at the information visit, signing of informed consent, and all study visits

Exclusion Criteria:

* Clinically relevant history of abnormal physical or mental health interfering with the study as determined by medical history taking and physical examinations obtained during the screening visit and/or at the study day as judged by the investigator;
* Clinically relevant abnormal laboratory results, electrocardiogram (ECG) and vital signs, or physical findings at screening and/or at the start of the study day (as judged by the investigator);
* Unwilling to or unable to stop smoking on the study day until the end of the study day
* Other causes that can explain cognitive symptoms including but not limited to: delirium, multiple sclerosis, amyotrophic lateral sclerosis, progressive supranuclear palsy, mental retardation, infectious encephalitis that led to persistent cognitive deficits or head trauma with loss of consciousness that led to persistent cognitive deficits
* Use of neuroleptics
* Use of celiprolol or sotalol
* Use of MAO-A/B inhibitors
* Current use of centrally acting anticholinergics (e.g. oxybutynin, mebeverine, ipratropium(bromide))
* Use of benzodiazepine within 48 hours before a study day
* Current use of a CEI (rivastigmine, galantamine, donepezil)
* Alcohol abuse (defined as use of alcohol despite significant areas of dysfunction, evidence of physical dependence, and/or related hardship due to alcohol)
* Use of recreational drugs
* Concomitant use of inhibitors of CYP2D6 (a/o kinidine, paroxetine, fluoxetine) or of CYP3A4 (a/o ketoconazole, ritonavir); unless patients are on a stable dose without any recent or upcoming changes
* Any other condition that in the opinion of the investigator would complicate or compromise the study, or the well being of the subject.
* Any contra-indication for MRI

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-02; Primary Completion 2016-12 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Change on performance on executive function and on memory after active challenge | timepoints 1 hour, 2.5 hours and 3.5 hours
  Patients will perform multiple Neurocart tests: eye movement recording, pharmaco-EEG's, visual verbal language test (VVLT), Adaptive Tracker, Facial Recognition taks, N-back and Stop Signal test of which the Adaptive Tracker and VVLT have the main focus.

SECONDARY OUTCOMES:
Change on performance on other Neurocart tests after active challenge | Timepoints 1.0 hour, 2.5 hours and 3.5 hours
  Change of performance on the other tests: N-back, Facial recognition task, Stop Signal task, eye movements and pharmaco-EEG

OTHER OUTCOMES:
Locations and number of cerebrovascular lesions | Single MRI scan after screening
  If patients are suitable for the study and have signed the informed consent they will undergo a MRI (structural, DTI and RS-fMRI). Visual assessment of structural cerebrovascular lesions in each patients
Structural connectivity of white matter tracts | Single MRI after screening
  If patients are suitable for the study and have signed the informed consent they will undergo a MRI (structural, DTI and RS-fMRI). Assessment of structural connectivity of specific white matter tracts, known to be part of the cholinergic and monoaminergic system with FLS software
Functional connectivity in resting state networks | Single MRI, after screening
  If patients are suitable for the study and have signed the informed consent they will undergo a MRI (structural, DTI and RS-fMRI). Assessment functional connectivity in specific resting state networks
Maximum concentration (Cmax) | t-1.5, t=1, t=2.5, t=3.5
Time of Cmax (Tmax) | t=-1.5, t=1, t=2.5, t=3.5
Area under the Curve | t=-1.5, t=1, t=2.5,t=3.5

CONTACTS AND LOCATIONS:
Overall Officials: Niels D Prins, MD, PhD, Principal Investigator — VUmc
Locations (1):
- VU University Medical Center, Amsterdam, Netherlands

REFERENCES:
- [Derived] Leijenaar JF, Groeneveld GJ, Klaassen ES, Leeuwis AE, Scheltens P, Weinstein HC, van Gerven JMA, Barkhof F, van der Flier WM, Prins ND. Methylphenidate and galantamine in patients with vascular cognitive impairment-the proof-of-principle study STREAM-VCI. Alzheimers Res Ther. 2020 Jan 7;12(1):10. doi: 10.1186/s13195-019-0567-z. PMID 31910895
- [Derived] Leijenaar JF, Groeneveld GJ, van der Flier WM, Scheltens P, Klaassen ES, Weinstein HC, Biessels GJ, Barkhof F, Prins ND. Symptomatic Treatment of Vascular Cognitive Impairment (STREAM-VCI): Protocol for a Cross-Over Trial. JMIR Res Protoc. 2018 Mar 20;7(3):e80. doi: 10.2196/resprot.9192. PMID 29559423